CLINICAL TRIAL: NCT07064499
Title: CGM Boosted by Artificial Intelligence for Better Glycaemic Control in T2 Diabetes: a Real-life Multicentre Observational Study in Belgium.
Brief Title: CGM Boosted by Artificial Intelligence for Better Glycaemic Control in T2 Diabetes
Acronym: MAGIC-T2D
Status: Active, not recruiting | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2021470
Record Dates: First submitted 2025-07-11; First posted 2025-07-14 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
Keywords: Evolution of Type 2 Diabetes Following CGM Introduction; Progression of Type 2 Diabetes Across Endotypes Following CGM Initiation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Title: CGM Boosted by Artificial Intelligence for better glycaemic control in T2 Diabetes : a real-life multicenter observational study in Belgium - MAGIC-T2D

Background: In Belgium, since May 2023, reimbursement for continuous glucose monitoring systems has been extended to people with type 2 diabetes taking multiple injections of insulin. Despite the results of previous studies, the impact of this technology in terms of glycaemic control and patient-reported outcomes (PROMs) in real life for patients with type 2 diabetes is still unclear.

Objective: To evaluate the impact of the CGMs on glycemic control and PROMs in people living with type 2 diabetes under real-life conditions.

Methods and analysis: In a multicenter real-world observational study, more than 440 people with type 2 diabetes under multiple daily injection therapy who start to be monitored by a CGM in one of the 13 participating Belgian centers, will be followed for a period of 24 months.

Outcomes: The primary and secondary endpoint are respectively the evolution of time spent in range (defined as a sensor glucose value between 70 and 180 mg/dL) and HbA1c from before start to 12 months after start of the CGM.

Exploratory objectives will be studied using artificial intelligence (AI) to study glucose profiles to characterize the heterogeneity of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes on MDI and starting CGM

Exclusion Criteria:

* Dialysis
* Treatment that raises blood sugar levels (corticosteroids, etc.)
* Secondary and type 1 diabetes
* Patient not able to sign the Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with type 2 diabetes on multiple insulin injections, monitored in the endocrinology-diabetology departments of participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of TIR (glucose 70-180 mg/dl) over a 12-month period after initiation of CGM in patients with T2D treated with MDI regimens. | From registration to end of 1-year follow-up

SECONDARY OUTCOMES:
Evolution of Hba1c over a 12-month period after initiation of CGM | From registration to end of 1-year follow-up

OTHER OUTCOMES:
Evolution of TIR according to T2D endotypes as defined by Ahlqvist et al. | From registration to end of 1-year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- HUB-Hôpital ERASME, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of data only after assessment of the request by our Ethics Committee and the Clinical Trials Centre of the HUB-Hôpital Erasme

REFERENCES:
- [Background] Zaccardi F, Khunti K. Glucose dysregulation phenotypes - time to improve outcomes. Nat Rev Endocrinol. 2018 Nov;14(11):632-633. doi: 10.1038/s41574-018-0092-3. No abstract available. PMID 30202117
- [Background] Hall H, Perelman D, Breschi A, Limcaoco P, Kellogg R, McLaughlin T, Snyder M. Glucotypes reveal new patterns of glucose dysregulation. PLoS Biol. 2018 Jul 24;16(7):e2005143. doi: 10.1371/journal.pbio.2005143. eCollection 2018 Jul. PMID 30040822
- [Background] Slieker RC, Donnelly LA, Fitipaldi H, Bouland GA, Giordano GN, Akerlund M, Gerl MJ, Ahlqvist E, Ali A, Dragan I, Festa A, Hansen MK, Mansour Aly D, Kim M, Kuznetsov D, Mehl F, Klose C, Simons K, Pavo I, Pullen TJ, Suvitaival T, Wretlind A, Rossing P, Lyssenko V, Legido-Quigley C, Groop L, Thorens B, Franks PW, Ibberson M, Rutter GA, Beulens JWJ, 't Hart LM, Pearson ER. Replication and cross-validation of type 2 diabetes subtypes based on clinical variables: an IMI-RHAPSODY study. Diabetologia. 2021 Sep;64(9):1982-1989. doi: 10.1007/s00125-021-05490-8. Epub 2021 Jun 10. PMID 34110439
- [Background] Ahlqvist E, Storm P, Karajamaki A, Martinell M, Dorkhan M, Carlsson A, Vikman P, Prasad RB, Aly DM, Almgren P, Wessman Y, Shaat N, Spegel P, Mulder H, Lindholm E, Melander O, Hansson O, Malmqvist U, Lernmark A, Lahti K, Forsen T, Tuomi T, Rosengren AH, Groop L. Novel subgroups of adult-onset diabetes and their association with outcomes: a data-driven cluster analysis of six variables. Lancet Diabetes Endocrinol. 2018 May;6(5):361-369. doi: 10.1016/S2213-8587(18)30051-2. Epub 2018 Mar 5. PMID 29503172
- [Background] Haak T, Hanaire H, Ajjan R, Hermanns N, Riveline JP, Rayman G. Flash Glucose-Sensing Technology as a Replacement for Blood Glucose Monitoring for the Management of Insulin-Treated Type 2 Diabetes: a Multicenter, Open-Label Randomized Controlled Trial. Diabetes Ther. 2017 Feb;8(1):55-73. doi: 10.1007/s13300-016-0223-6. Epub 2016 Dec 20. PMID 28000140
- [Background] McGill JB, Ahmann A. Continuous Glucose Monitoring with Multiple Daily Insulin Treatment: Outcome Studies. Diabetes Technol Ther. 2017 Jun;19(S3):S3-S12. doi: 10.1089/dia.2017.0090. PMID 28585875
- [Background] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185